CLINICAL TRIAL: NCT05944926
Title: Improving Outcomes in Depression in Primary Care in a Low Resource Setting
Acronym: OptimizeD
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Harvard Medical School (HMS and HSDM) (Other)
Collaborators: Sangath (Other); All India Institute of Medical Sciences, Bhopal (Other); Vanderbilt University (Other); Brigham and Women's Hospital (Other); Centre for Addiction and Mental Health (Other); Massachusetts General Hospital (Other); Harvard School of Public Health (HSPH) (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Vikram Patel, Co-Principal Investigator; The Pershing Square Professor of Global Health at Harvard Medical School, Harvard Medical School (HMS and HSDM)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB20-2144; CTRI/2024/01/061932 (Other: Clinical Trials Registry - India (ICMR-NIMS)); 1R01MH121632-01A1 (NIH)
Record Dates: First submitted 2023-06-02; First posted 2023-07-13 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Depression; Depressive Disorder
MeSH Terms: conditions — Depression; Depressive Disorder | interventions — Antidepressive Agents; Fluoxetine

STUDY DESIGN:
Intervention Model Description: Fluoxetine versus a contextually adapted version of behavioral activation called the Healthy Activity Program (HAP) delivered by non-specialists for treatment of depression
Who Masked: Outcomes Assessor
Masking Description: Masked (blinded) field-based assessors will conduct all outcome assessments
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Activity Program (HAP) (Experimental): HAP is a brief psychological treatment adapted from behavioral activation therapy, an empirically supported psychological treatment recommended by WHO.
  Interventions: Behavioral: Healthy Activity Program (HAP)
- Antidepressant medication (fluoxetine) (Experimental): Fluoxetine is a selective serotonin reuptake inhibitors (SSRIs) and one of the safest medications used to treat depression. It is a routinely used medication and part of the Essential Drug List (EDL) in India.
  Interventions: Drug: Antidepressant medication (fluoxetine)

INTERVENTIONS:
Behavioral: Healthy Activity Program (HAP) — HAP, delivered over 6-8 sessions by non-specialist healthcare workers, has behavioural activation as the core psychological strategy along with other strategies such as problem-solving and activation of social networks.
  Arms: Healthy Activity Program (HAP)
Drug: Antidepressant medication (fluoxetine) — Patients assigned to antidepressant medication will start on fluoxetine 20 mg/day and can be raised to 40 mg/day (the maximum mandated by treatment guidelines for primary care in India) at week 3 or 6 for patients who have yet to remit. Participants who do not tolerate fluoxetine can be switched to escitalopram at week 6 (10mg which can be titrated up to 20 mg).
  Arms: Antidepressant medication (fluoxetine)

SUMMARY:
The OptimizeD study aims to improve outcomes in depression in primary care in India. This study will randomize 1500 patients with moderate to severe depression to either psychotherapy based on behavioral activation called the Healthy Activity Program (HAP) or antidepressant medication (fluoxetine).

The study has two primary objectives:

1. Use patient characteristics to generate a precision treatment rule based on baseline information for predicting in advance what works best for whom (and which patients are unlikely to respond to either treatment and should be referred to specialist care).
2. Conduct a cost-effectiveness analysis by comparing relative costs and effectiveness between those who were randomly allocated to their optimal treatment with those who were randomly allocated to a non-optimal treatment based on the precision treatment rule.

DETAILED DESCRIPTION:
Depression is the leading mental health contributor to the Global Burden of Disease. The World Health Organization's mhGAP initiative advocates the use of brief psychological therapies such as behavioral activation or antidepressant medications as first-line options for the treatment of moderate to severe depression in primary care settings, but not all patients will fully remit on either treatment. It is likely that different patients will respond to different treatments, but the optimal treatment for each individual remains unknown (and which patients are unlikely to respond to either treatment and should be referred to specialist care). Enhancing our ability to determine the optimal intervention for a particular patient has the potential to enhance the overall effectiveness of mental health care delivery in a more cost-efficient manner. This is a critical gap in knowledge in the treatment of depression across clinical settings globally.

The main objective of the OptimizeD study is to determine whether different patients respond differentially to brief psychological treatment or a widely used generic SSRI and, if so, whether one can optimize outcomes in a cost-effective fashion for primary care patients with moderate to severe depression.

The study has two specific aims and two exploratory aims:

* Specific Aim 1 (Clinical and Functional Outcomes): To evaluate the effectiveness of optimization via generating a precision treatment rule (PTR) on patients with moderate to severe depression randomized to either psychotherapy based on behavioral activation called the Healthy Activity Program (HAP) or antidepressant medication (fluoxetine). The study will use machine learning to develop the PTR, using a wide range of clinical, socio-economic, and neuro-cognitive characteristics measured at baseline as predictors. The investigators hypothesize that patients randomized by chance to their optimal intervention will be more likely to remit and recover than patients who are not.
* Specific Aim 2 (Cost-effectiveness Outcomes): To assess the costs of optimal vs. non-optimal treatments and to conduct a cost-effectiveness analysis by comparing relative costs and effectiveness between those who were randomly allocated to their optimal treatment with those who were randomly allocated to a non-optimal treatment, based on the PTR developed in Aim 1. The investigators hypothesize that optimizing will be more cost-effective than not.
* Exploratory Aim 1 (Mediators): To explore whether one can use the PTR to make our tests of mediation more precise. Patients who respond differentially to different treatments adhere to different causal mechanisms, and inclusion of the PTR in interaction terms with the purported mediators should facilitate the detection of moderated mediation among patients who show specificity of response. The investigators will also consider whether treatment-related factors (e.g., adherence, quality) act as mediators of the effects of each treatment on remission and recovery. This exploratory aim will offer insights into mechanisms of action for each treatment.
* Exploratory Aim 2 (Genetic Predictors): To explore whether polygenic risk scores and other biomarkers can enhance the prediction of both general and differential response to either treatment.

As a secondary objective, the study will evaluate the effectiveness of optimization in the long-term. The investigators hypothesize that patients allocated to their optimized treatment will be more likely to recover than patients who are allocated to their non-optimal treatment.

All trial procedures used in the main trial were first evaluated in a pilot study (NCT06153004), which employed the same design and methods to assess feasibility across recruitment, randomization, retention, treatment adherence and fidelity, and data quality assurance.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be adults aged 18 or over of any gender attending one of the selected Primary Health Care Centers with a "diagnosis" of moderate to severe depression based on scores of 10 or above on the Patient Health Questionnaire-9 (PHQ-9).

Exclusion Criteria:

1. Women who are pregnant or are breastfeeding or lactating
2. Patients with a history of psychosis, including schizophrenia spectrum disorders or bipolar disorder.
3. Participants planning to permanently move out of the study area during the follow-up period.
4. Patients with evidence of cognitive impairment.
5. Patients who do not speak either English or Hindi.
6. Patients who are undergoing treatment for depression at the time of recruitment or who completed treatment within one month prior to recruitment
7. Patients at imminent risk for suicide
8. Patients from households in which another member has been recruited into the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2024-03-18 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Depression remission | 3 months post recruitment
  Remission is defined as PHQ-9 total score < 5. The PHQ-9 is a self-report measure of depressive symptoms in the prior 2 weeks. Items are rated on a 4-point Likert scale from 0 (not at all) to 3 (nearly every day), with total scores ranging from 0 to 27, where higher scores indicate more severe depressive symptoms. We will dichotomised the total score using the cut-off score of 5.

SECONDARY OUTCOMES:
Cost-effectiveness of optimization | 3-, 6-, 9-, 12-months post recruitment
  Cost-effectiveness analysis by comparing costs and effectiveness between those who were randomly allocated to their optimal treatment vs. those who were randomly allocated to a non-optimal treatment. Effectiveness will be measures by (1) likelihood of remission and (2) Quality Adjusted Life Years (QALYs). Costs of treatments include three components: system-level costs incurred at the health facility level, individual costs incurred by HAP counselors and Medical Officers in delivering each treatment, and costs incurred by patients for participating in the treatment. See section below for a description of these measures.
Depression severity, as measured by the Patient Health Questionnaire-9 (PHQ-9) | 3-, 6-, 9-, 12-months post recruitment
  The PHQ-9 is a 9-item self-report scale to screen for symptoms of depression. Items are rated on a 4-point Likert scale from 0 (not at all) to 3 (nearly every day), with total scores ranging from 0 to 27, where higher scores indicate more severe depressive symptoms.
Generalized Anxiety Disorder Assessment (GAD-7) | 3-, 6-, 9-, 12-months post recruitment
  The GAD-7 is a 7-item self-report scale to screen for symptoms of generalized anxiety disorder. Items are rated on a 4-point Likert scale from 0 (not at all) to 3 (nearly every day), with total scores ranging from 0 to 21, where higher scores indicate more severe anxiety symptoms.
WHO Disability Assessment Schedule II (WHODAS-II) | 3-, 6-, 9-, 12-months post recruitment
  The WHODAS-II consists of 12-items that capture level of functioning across six life domains including cognition, mobility, self-care, getting along, life activities, and participation in society. Each item ranges from 1 (none) to 5 (extreme), with total scores from 12-60. Raw scores are then converted to a summary score ranging from 0 (no disability) to 100 (full disability).
Minimal Clinically Important Difference (MCID) | 3-, 6-, 9-, 12-months post recruitment
  We will use the anchor-based approach for estimating MCID that ties change in outcome on the PHQ-9 to the patient's subjective sense of improvement. We will follow Weobong (2017) methodology to compute this.
World Health Organization Well-Being Index (WHO-5) | 3-, 6-, 9-, 12-months post recruitment
  The WHO-5 consists of 5-items that measure current mental well-being. Each item is rated on 6-point Likert scale, ranging from 0 (at no the time) to 5 (all of the time). The total raw score, ranging from 0 to 25, is multiplied by 4 to give the final score, with 0 representing the worst imaginable well-being and 100 representing the best imaginable well-being.

OTHER OUTCOMES:
Recovery from depression as measured by the PHQ-9 | 12-month post recruitment
  Recovery from depression symptoms is defined as going nine months without relapse (PHQ-9 ≥5) following remission.
Client Service Receipt Inventory (CSRI) | 3-, 6-, 9-, 12-months post recruitment
  Out-of-pocket costs for receiving care and the related non-medical costs.
Quality Adjusted Life Years (QALYs) as measured by WHODAS II | 3-, 6-, 9-, 12-months post recruitment
  WHODAS II is a 12-item scale that captures the level of functioning across six life domains, including cognition, mobility, self-care, getting along, life activities, and participation in society (Saltychev et al., 2021). Each item ranges from 1 (none) to 5 (extreme), with total simple scores from 12-60. Standardized summary scores will be converted to a preference-weighted utility index, which will then be used to compute the additional number of QALYs generated by the interventions. The answers to two questions in WHODAS can be used to estimate the number of days in the previous month that someone was completely unable to work or able to work only part time because of a health condition.

CONTACTS AND LOCATIONS:
Overall Officials: Vikram Patel, MD, Principal Investigator — Vikram_Patel@hms.harvard.edu
Locations (1):
- Sangath, Bhopal, Madhya Pradesh, India

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared through the NIMH Data Archive. To ensure participant privacy and data security, all shared data will be de-identified according to established protocols and guidelines. The data sharing plan will be periodically reviewed and updated, as necessary, to align with evolving best practices, policies, and guidelines for data sharing.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available indefinitely or for as long as the NIMH repositories support it.
Access Criteria: Researchers and interested parties who wish to access the data can submit a formal data access request to the NIMH Data Archive. Researchers who gain access to the data will be required to comply with the data usage policies and guidelines set forth by the NIMH Data Archive.
URL: https://nda.nih.gov/

REFERENCES:
- [Background] Weobong B, Weiss HA, McDaid D, Singla DR, Hollon SD, Nadkarni A, Park AL, Bhat B, Katti B, Anand A, Dimidjian S, Araya R, King M, Vijayakumar L, Wilson GT, Velleman R, Kirkwood BR, Fairburn CG, Patel V. Sustained effectiveness and cost-effectiveness of the Healthy Activity Programme, a brief psychological treatment for depression delivered by lay counsellors in primary care: 12-month follow-up of a randomised controlled trial. PLoS Med. 2017 Sep 12;14(9):e1002385. doi: 10.1371/journal.pmed.1002385. eCollection 2017 Sep. PMID 28898283
- [Derived] Pozuelo JR, Lahiri A, Singh RSP, Kushwah A, Khanduri M, Shukla A, Khan A, G S, Shende V, Parashar Y, Mehra YK, Bhan A, Kessler RC, Singla DR, Naslund JA, Choi KW, Cuijpers P, DeRubeis R, Herzallah MM, Lu C, Smoller JW, VanderWeele TJ, Rozatkar AR, Modak T, Joel MM, Biswas D, Atal S, Kulsum U, Hollon SD, Patel V. Optimizing treatment for depression in primary care using psychotherapy versus antidepressant medication in a low-resource setting: protocol for the OptimizeD randomized controlled trial. BMC Psychiatry. 2025 Jul 30;25(1):744. doi: 10.1186/s12888-025-07030-9. PMID 40739549
- [Derived] Pozuelo JR, Lahiri A, Singh RSP, Kushwah A, Khanduri M, Shukla A, Khan A, G S, Shende V, Parashar Y, Mehra YK, Bhan A, Kessler RC, Singla DR, Naslund JA, Choi K, Cuijpers P, DeRubeis R, Herzallah M, Lu C, Smoller JW, VanderWeele TJ, Rozatkar A, Joel MM, Biswas D, Atal S, Kulsum U, Hollon SD, Patel V. Optimizing Treatment for Depression in Primary Care Using Psychotherapy Versus Antidepressant Medication in a Low-Resource Setting: Protocol for the OptimizeD Randomized Controlled Trial. Res Sq [Preprint]. 2025 May 23:rs.3.rs-6716211. doi: 10.21203/rs.3.rs-6716211/v1. PMID 40470239
- See also: Study overview — https://mentalhealthforalllab.hms.harvard.edu/optimized